CLINICAL TRIAL: NCT03155659
Title: Fish, Polyunsaturated Fatty Acids Intake and Mortality: Analysis of CHNS and NHANES
Brief Title: Fish, Polyunsaturated Fatty Acids Intake and Mortality
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: National Institute of Health and Nutrition (Other Government)
Responsible Party: Principal Investigator, Jingjing Jiao, Associate Professor, Zhejiang University
Other Study IDs: Cohort_PUFA
Record Dates: First submitted 2017-05-13; First posted 2017-05-16 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Polyunsaturated Fatty Acids; Mortality
Keywords: Fish; Polyunsaturated fatty acids; Mortality; CHNS; NHANES

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Data linking fish, polyunsaturated fatty acids intake and mortality are lacking and conflicting. We aim to use data from the China Health and Nutrition Survey (CHNS) and National Health and Nutrition Examination Survey (NHANES) to investigate the associations of fish and polyunsaturated fatty acids (PUFA) intake with mortality in Chinese and US populations. The study findings will be informative for addressing the role of fish and specific PUFA in human health and improve basis for dietary recommendations.

DETAILED DESCRIPTION:
Data from the China Health and Nutrition Survey (CHNS, from 1989 to 2011) and National Health and Nutrition Examination Survey (NHANES), including NHANES III conducted in 1988-1994 and continuous NHANES 1999-2010 were used to investigate the associations of fish and polyunsaturated fatty acids intake with mortality.The following variables were used:

1. Demographics: age, sex, race/ethnicity, residence
2. Socioeconomic variables: education, marital status,
3. Dietary variables: Intakes of fish, polyunsaturated fatty acids, total energy, vegetables, fruits, red meat and saturated fat
4. Clinical assessments: hypertension, diabetes, cancer, cardiovascular disease (CVD), family history of CVD

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥20 with complete data on diet and follow-up time

Exclusion Criteria:

* Missing information for mortality
* Cardiovascular disease
* Cancer

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CHNS is an ongoing, large-scale, household-based cohort starting in 1989. The survey used a multi-stage, random cluster process to draw a sample of 9 provinces and municipal cities, which take up about half of Chinese population. NHANES is also a nationally-representative study of nutrition and health for individuals residing in the U.S. Our study included participants in CHNS and NHANES who met the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 50145 (Actual)
Dates: Start 1989-01 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Total Mortality | From baseline until death or censoring on 31 December 2011, whichever came first, assessed up to an average of 10 years
  Total Mortality from All Causes

SECONDARY OUTCOMES:
Cause-specific mortality | From baseline until death or censoring on 31 December 2011, whichever came first, assessed up to an average of 10 years
  Cause-specific mortality from diseases

REFERENCES:
- [Result] Zhao LG, Sun JW, Yang Y, Ma X, Wang YY, Xiang YB. Fish consumption and all-cause mortality: a meta-analysis of cohort studies. Eur J Clin Nutr. 2016 Feb;70(2):155-61. doi: 10.1038/ejcn.2015.72. Epub 2015 May 13. PMID 25969396
- [Result] Rizos EC, Ntzani EE, Bika E, Kostapanos MS, Elisaf MS. Association between omega-3 fatty acid supplementation and risk of major cardiovascular disease events: a systematic review and meta-analysis. JAMA. 2012 Sep 12;308(10):1024-33. doi: 10.1001/2012.jama.11374. PMID 22968891
- [Derived] Zhuang P, Wang W, Wang J, Zhang Y, Jiao J. Polyunsaturated fatty acids intake, omega-6/omega-3 ratio and mortality: Findings from two independent nationwide cohorts. Clin Nutr. 2019 Apr;38(2):848-855. doi: 10.1016/j.clnu.2018.02.019. Epub 2018 Mar 3. PMID 29551407
- See also: Related Info — http://dx.doi.org/10.1038/ejcn.2015.72